CLINICAL TRIAL: NCT05288491
Title: Concordance Study of CD30 Expression Detected by Multiple Immunohistochemistry Assays and VENTANA CD30 Assay in Chinese Lymphoma Patients
Brief Title: A Study of Chinese Adults With Lymphoma
Acronym: CREDIT
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C25025
Record Dates: First submitted 2022-03-15; First posted 2022-03-21 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Malignant Lymphoma: All participants diagnosed with histopathologically confirmed malignant lymphoma will be enrolled and observed retrospectively. Complete medical information will be collected at the time of enrollment via chart review.

SUMMARY:
The main aim of this study is to improve methods of clinical testing and therapy for lymphoma participants.

This study will involve collecting information about participants from past medical records.

DETAILED DESCRIPTION:
This is an observational, non-interventional, retrospective study to evaluate staining and interpretation concordance of CD30 expression detected by 9 immunohistochemistry (IHC) assays and VENTANA CD30 IHC assay in Chinese lymphoma participants.

This study will enroll approximately 1000 participants. The data will be collected via chart review in the electronic case report forms (eCRFs). All the participants will be assigned to a single observational cohort:

• Participants With Malignant Lymphoma

This multi-center trial will be conducted in China. The overall duration of the study will be approximately 21 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with diagnosis of cHL, ALCL, MF-LCT, DLBCL, PMBL, ENKTCL, PTCL-NOS, AITL and PCCD30+TCLPD.
2. Participants with available FFPE samples archived within 3 years.
3. Whose tissue slides of FFPE samples were previously IHC stained, their CD30 expression showed as well-localized positive stain and investigator deemed appropriate for evaluation.

Exclusion Criteria:

1. Sample is not sufficient for CD30 testing.
2. Incomplete sample information including key demographic characteristic, clinicopathological parameters and previous CD30 testing results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese participants who have histopathologically confirmed or diagnosed with malignant lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 934 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Positive Cells for CD30 Expression Detected by 9 IHC Assays and VENTANA CD30 Assay | Up to 12 months
  VENTANA CD30 assay (Ber-H2 (Ventana, Roche) + Ventana BenchMark) is standardized method preset in this study. The tissue slides from one Formalin-fixed and Paraffin-embedded (FFPE) samples will be stained by VENTANA CD30 IHC assay and at least one selected IHC assay. The staining concordance of percentage of CD30 positive cells for CD30 expression detected by 9 IHC assays and VENTANA CD30 assay will be respectively evaluated by intraclass correlation coefficient (ICC), Bland-Altman and Pearson correlation method. The selected 9 IHC assays will be used for evaluation of samples are: 1) umAB256 (Zhongshanjinqiao) + Ventana BenchMark, 2) Ber-H2 (Maixin) + Ventana BenchMark, 3) Ber-H2 (Maixin) + DAKO, 4) Ber-H2 (DAKO) + DAKO, 5) Ber-H2 (DAKO) + Ventana BenchMark, 6) umAB256 (Zhongshanjinqiao) + Leica, 7) JCM182 (Leica) + Ventana BenchMark, 8) JCM182 (Leica) + Leica, 9) Ber-H2 (DAKO) + Leica.

SECONDARY OUTCOMES:
Percentage of Positive Cells for CD30 Expression Detected by IHC Assays and Interpreted by Pathologists | Up to 12 months
  The tissue slides from one FFPE samples will be stained by VENTANA CD30 IHC assay and at least one selected IHC assay. CD30 expression of all immunostained slides will be independently interpreted as a percentage of CD30 positive cells by trained pathologists at sites. The interpreting concordance of pathologists at sites and the expert panel by assessing CD30 expression detected by various IHC assays will be also evaluated by ICC, Bland-Altman and Pearson correlation method.
Percentage of Participants With Different Lymphoma Subtypes | Up to 12 months
  The distribution of CD30 expression in Chinese lymphoma participants will be evaluated by percentage of Chinese participants with different lymphoma subtypes. Samples from participants with diagnosis of 9 lymphoma subtypes: Classical hodgkin's lymphoma (cHL), anaplastic large cell lymphoma (ALCL), large cell transformation of mycosis fungoides (MF-LCT), diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBL), extranodel nature killer or T cell lymphoma (ENKTCL), peripheral T cell lymphoma, not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL) and primary cutaneous CD30-positive lymphoproliferative disorders (PCCD30+TCLPD) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- China (19):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Medical College of Hust, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/